CLINICAL TRIAL: NCT05435521
Title: MOVIhNG Study: Impact of a Personalized Multicomponent Exercise Program in Real Conditions on Physical Function, Frailty, and Quality of Life Among Older Adults With HIV
Brief Title: Impact of a Personalized Multicomponent Exercise Program in Real Conditions Among Older Adults With HIV
Acronym: MOVIhNG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Universitario Ramon y Cajal (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Matilde Sánchez Conde, Principal Investigator, Hospital Universitario Ramon y Cajal
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI20/01078
Record Dates: First submitted 2022-06-13; First posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Frailty; Quality of Life; Physical Inactivity; Body Composition
Keywords: HIV; Frailty; Exercise; Physical function; Quality of life
MeSH Terms: conditions — Frailty; Sedentary Behavior; Motor Activity | interventions — Pliability; Body Composition

STUDY DESIGN:
Intervention Model Description: Multicentric prospective longitudinal clinical study with intervention with a control group (Non HIV patients) and a group wih HIV
Masking Description: Masking will not be performed due to the necessity of active supervision and follow up of the activity program
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- People living with HIV group 40 participants (Experimental): 40 participants with HIV
  Interventions: Behavioral: Personalized multicomponent exercise program (strength, resistance, balance, and flexibility) (PMEP); Other: Body composition; Other: Musculoskeletal and visceral Ultrasound
- People without HIV (Active Comparator): 20 participants without HIV
  Interventions: Behavioral: Personalized multicomponent exercise program (strength, resistance, balance, and flexibility) (PMEP); Other: Body composition; Other: Musculoskeletal and visceral Ultrasound

INTERVENTIONS:
Behavioral: Personalized multicomponent exercise program (strength, resistance, balance, and flexibility) (PMEP) — Physical activity expert will design for each participant a personalized exercise program according to baseline situation and previous physical activity. Both will be measured prior to initiation of activity program. Each participant is free to perform physical activity program at his house, outdoor or in a gym as long as it fulfills the prespecified requirements. Exercise programs will be acquired a more personalized shape during the course of the study.
  In order to motivate participants, personal motivational messages will be sent each week through mail contact or using "WhatsApp" Social Media.
  Physical activity will be registered in an activity wristband delivered to each participant at baseline evaluation.
Other: Body composition — Analyze the effects of PMEP on body composition in each evaluation using an impedance threshold device
Other: Musculoskeletal and visceral Ultrasound — Quadriceps muscle ultrasound (US) of the rectus femoris measured in each evaluation in order to analyze the effects of PMEP Visceral fat will be analyzed in each visit

SUMMARY:
Longitudinal prospective multicenter study with intervention and control groups and a two-year follow up. Participants will include 40 sedentary adults 50 years old or older with HIV infection and 20 sedentary adults 50 years old or older without HIV infection. Our main objective is to analyze the effects of a personalized multicomponent exercise program (strength, resistance, balance, and flexibility) (PMEP) on physical function, frailty, and quality of life among older adults with HIV. As secondary objectives, we are going to analyze the effects of a PMEP on body composition, muscle function biomarkers, immunological biomarkers, microbiome, and adherence to PMEP in real conditions under intense, moderate nonexistent monitoring.

DETAILED DESCRIPTION:
PMEPs will be designed according to the specific characteristics of each participant and their grade of usual physical activity. Physical activity will be registered on physical activity bracelets to get objective information in order to evaluate adherence to the PMEP. A global evaluation of the patients will be made at baseline and months 3, 6, and 12. At each evaluation, samples of blood, stool, urine, and saliva will be taken, and a phone meeting will be scheduled at month 24.

ELIGIBILITY:
Inclusion Criteria:

* People living with HIV (Control group not included)
* Age equal or older to 50 years old at initiation of study
* Sedentary individuals: < 150 minutes per week of moderate physical activity.
* Absence of physical limitations which impede the performance of a light or moderate physical activity program

Exclusion Criteria:

* Individuals with one or more of the following diseases:

* Acute myocardial infarction (in the previous 3-6 months) or unstable angina
* Uncontrolled cardiac arrythmias
* Severe aortic stenosis
* Acute Pericarditis/ Endocarditis
* Poorly controlled high blood pressure (> 180/100 mmHg)
* Acute thromboembolic disease
* Acute severe cardiac heart failure

Ages: 50 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Effects of a personalized multicomponent exercise program (strength, resistance, balance, and flexibility) (PMEP) | 12 months
  To analyze the effects of a personalized multicomponent exercise program (strength, resistance, balance, and flexibility) (PMEP) on physical function among older adults with HIV.
  Physical function will be assessed using Short Physical Performance Battery" (SPPB or Guralnik test) will be measured in each evaluation
Effects of a personalized multicomponent exercise program (strength, resistance, balance, and flexibility) (PMEP) | 12 months
  To analyze the effects of a personalized multicomponent exercise program (strength, resistance, balance, and flexibility) (PMEP) on frailty among older adults with HIV.
  Frailty will be assessed using Fried phenotype in each visit
Effects of a personalized multicomponent exercise program (strength, resistance, balance, and flexibility) (PMEP) | 12 months
  To analyze the effects of a personalized multicomponent exercise program (strength, resistance, balance, and flexibility) (PMEP) on quality of life among older adults with HIV.
  Quality of life will be assessed using World Health Organization Quality of Life HIV instrument (WHOQOL-HIV-BREF)

SECONDARY OUTCOMES:
Comparison of PMEP effects between HIV and non HIV participants of the same age | 12 months
  In order to measure if the impact of PEMP in older adults with HIV is higher than in non HIV participants, 20 individuals of similar age have been included without HIV infection.
  Impact of PMEP will be measured analyzing frailty which will be assessed using Fried phenotype in each visit
Comparison of PMEP effects between HIV and non HIV participants of the same age | 12 months
  In order to measure if the impact of PEMP in older adults with HIV is higher than in non HIV participants, 20 individuals of similar age have been included without HIV infection.
  Impact of PMEP will be measured using the Short Physical Performance Battery" (SPPB or Guralnik test) which will be measured in each evaluation
Comparison of PMEP effects between HIV and non HIV participants of the same age | 12 months
  In order to measure if the impact of PEMP in older adults with HIV is higher than in non HIV participants, 20 individuals of similar age have been included without HIV infection.
  Impact of PMEP will be measured analyzing body composition (BMI) in kg/m^2 which will be measured in each evaluation in order to assess changes throughout study period
Comparison of PMEP effects between HIV and non HIV participants of the same age | 12 months
  In order to measure if the impact of PEMP in older adults with HIV is higher than in non HIV participants, 20 individuals of similar age have been included without HIV infection.
  Impact of PMEP will be measured with Rectus femoris in cm measurements of both legs and visceral fat measurements in cm will be performed using ultrasound in each evaluation in order to see evolution in these parameters
Assesment of body composition evolution after implementation of PMEP using a segmental multi frequency body composition analyser though electrical impedance | 12 months
  Electrical bioimpedance measurement wil be performed in baseline evaluation and 3, 6 and 12 months after initiation of PMEP.
  The device used is Tanita MC-780 S MA analyzing BMI in kg/m^2
Effects of PMEP in muscular and immunological biomarkers and in microbiome | 12 months
  At each evaluation (baseline, 3, 6 and 12 months), samples of blood, stool, urine, and saliva will be taken. Immunosenescence and chronic inflammation in HIV are considered at the present moment one of the main drivers of non AIDS comorbidities. Several studies have shown solid conclusions positioning physical activity as a clear intervention which reduces chronic inflammation in individuals without HIV as well as in people living with HIV.
Evaluation of PMEP adherence | 12 months
  PMEP adherence rate will be assessed in real life conditions with different supervision levels (narrow, medium and no supervision at all)

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available via the Clinical Study Data Request site (currently under development)
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Branas F, Diaz-Alvarez J, Fernandez-Luna J, Vasquez-Brolen BD, Garcia-Molina R, Moreno E, Ryan P, Martinez-Sanz J, Luna L, Martinez M, Dronda F, Sanchez-Conde M. A 12-week multicomponent exercise program enhances frailty by increasing robustness, improves physical performance, and preserves muscle mass in older adults with HIV: MOVIhNG study. Front Public Health. 2024 Apr 17;12:1373910. doi: 10.3389/fpubh.2024.1373910. eCollection 2024. PMID 38694984